CLINICAL TRIAL: NCT00466999
Title: Sublingual Misoprostol Versus Standard Surgical Care for the Treatment of Incomplete Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2.2.2
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Incomplete Abortion
Keywords: misoprostol; incomplete abortion; PAC
MeSH Terms: conditions — Abortion, Incomplete | interventions — Misoprostol; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- surgery (Active Comparator): standard surgical treatment (either dilation and curettage or manual vacuum aspiration)
  Interventions: Procedure: surgery
- misoprostol (Active Comparator): 400 mcg misoprostol
  Interventions: Drug: misoprostol

INTERVENTIONS:
Drug: misoprostol — single dose of 400 mcg misoprostol administered sublingually
  Arms: misoprostol
Procedure: surgery — standard surgical treatment (dilation and curettage or manual vacuum aspiration)
  Arms: surgery

SUMMARY:
In this study, we will compare the safety and efficacy of 400 mcg sublingually administered misoprostol alone to standard surgical care for the treatment of incomplete abortion. This study will provide important data on the role of misoprostol in health services offering an array of treatments for incomplete abortion. Women could significantly benefit from a non-invasive treatment option for incomplete abortion. While safe surgical services are becoming more widespread, there is still a serious risk of complications from these procedures. Especially in developing countries, infection, hemorrhage and uterine damage are still too common. Medical treatment of incomplete abortion using misoprostol would be a tremendous step to reducing morbidity and mortality due to abortion complications.

ELIGIBILITY:
Inclusion Criteria:

* Uterine size no larger than 12 weeks LMP at time of presentation for care.
* Past or present history of vaginal bleeding during pregnancy.
* Open cervical os.
* If ultrasound used evidence of incomplete abortion with substantial debris in the uterus.
* All women would have been advised to have surgical evacuation of the uterus if misoprostol was not available.
* General good health.
* Willing to provide contact information for purposes of follow-up.
* Also in Egypt: 21 years of age or over or parental permission (there is no minimum age requirement in Niger, Mauritania and Senegal).

Exclusion Criteria:

* Contraindications to study drug
* Signs of severe infection, defined as at least one of the following: 1) foul smelling discharge, 2) fever > 38 degrees C , 3) uterine tenderness
* Hemodynamic disturbances (pulse >110/min and systolic bp <100)
* Have an IUD in place; (the IUD may be removed making the woman eligible)
* Suspected ectopic pregnancy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2007-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Complete abortion without recourse to surgical intervention. | follow up visit 7 days after initial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Rasha Dabash, MPH, Study Director — Gynuity Health Projects; Ayisha Diop, MPH, Study Director — Gynuity Health Projects
Locations (6):
- Dandé District Hospital/Ziniaré District Hospital, Dande/Ziniare, Burkina Faso
- Egypt (2):
  - El-Galaa Teaching Hospital, Cairo
  - Shatby Maternity Hospital/Alexandria University, Shatby, Alexandria
- Cheikh Zayed Hospital, Nouakchott, Mauritania
- Maternite Issaka Gazobi, Niamey, Niger
- Centre de Sante Le Roi Baudouin, Guédiawaye, Senegal

REFERENCES:
- [Derived] Ghosh J, Papadopoulou A, Devall AJ, Jeffery HC, Beeson LE, Do V, Price MJ, Tobias A, Tuncalp O, Lavelanet A, Gulmezoglu AM, Coomarasamy A, Gallos ID. Methods for managing miscarriage: a network meta-analysis. Cochrane Database Syst Rev. 2021 Jun 1;6(6):CD012602. doi: 10.1002/14651858.CD012602.pub2. PMID 34061352
- [Derived] Shochet T, Diop A, Gaye A, Nayama M, Sall AB, Bukola F, Blandine T, Abiola OM, Dao B, Olayinka O, Winikoff B. Sublingual misoprostol versus standard surgical care for treatment of incomplete abortion in five sub-Saharan African countries. BMC Pregnancy Childbirth. 2012 Nov 14;12:127. doi: 10.1186/1471-2393-12-127. PMID 23150927
- [Derived] Blandine T, Ouattara AZ, Coral A, Hassane C, Clotaire H, Dao B, Lankoande J, Diop A, Blum J. Sublingual [corrected] misoprostol as first-line care for incomplete abortion in Burkina Faso. Int J Gynaecol Obstet. 2012 Nov;119(2):166-9. doi: 10.1016/j.ijgo.2012.05.036. Epub 2012 Aug 28. PMID 22935621
- [Derived] Dabash R, Ramadan MC, Darwish E, Hassanein N, Blum J, Winikoff B. A randomized controlled trial of 400-mug sublingual misoprostol versus manual vacuum aspiration for the treatment of incomplete abortion in two Egyptian hospitals. Int J Gynaecol Obstet. 2010 Nov;111(2):131-5. doi: 10.1016/j.ijgo.2010.06.021. PMID 20801444
- See also: Related Info — http://www.gynuity.org